CLINICAL TRIAL: NCT03309657
Title: A Prospective Pharmacokinetic Evaluation of the Plasma and Cerebrospinal Fluid Concentrations of a Single Dose Ceftolozane/Tazobactam in Infected Critically Ill Patients With an Indwelling External Ventricular Drain
Brief Title: Pharmacokinetics of Ceftolozane/Tazobactam in Plasma and Cerebrospinal Fluid
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royal Brisbane and Women's Hospital (Other Government)
Collaborators: The University of Queensland (Other)
Responsible Party: Principal Investigator, Jason Roberts, Professor, Royal Brisbane and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HREC/17/QRBW/117
Record Dates: First submitted 2017-07-30; First posted 2017-10-13 (Actual); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — ceftolozane, tazobactam drug combination

STUDY DESIGN:
Intervention Model Description: Open label pharmacokinetic study where enrolled critically ill patients with infection receive a single dose of ceftolozane-tazobactam (in addition to other active therapy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ceftolozane Tazobactam (Experimental): Infected patients with external intraventricular drain will receive a single dose of Ceftolozane/ tazobactam (3000mg) over 1 hour and will undergo blood , csf and urine sampling at specific times over an 8 hour period.
  Interventions: Drug: Ceftolozane/tazobactam

INTERVENTIONS:
Drug: Ceftolozane/tazobactam — This is an observational pharmacokinetic study whereby patients received a single dose of ceftolozane/tazobactam and plasma and cerebrospinal fluid samples were subsequently collected and analyzed to described the pharmacokinetics.
  Other Names: ZERBAXA

SUMMARY:
Ceftolozane/tazobactam is an emerging newly available antibiotic that has a broad spectrum of activity, and could be potentially useful in the management of central nervous system infections. However, data relating to penetration of ceftolozane/ tazobactam into the central nervous system, where a barrier against drug distribution exists (i.e. blood brain barrier), is currently limited. In critically ill patients this is all the more challenging as achieving adequate antibiotic concentrations even in blood is difficult.

The aim of this study is to describe the concentrations achieved in the cerebrospinal fluid (i.e. bodily fluid found surrounding and inside of the brain) and blood after a single dose of ceftolozane/tazobactam administered in critically ill patients with an existing external ventricular drain (i.e. a device used in neurosurgery that relieves elevated intracranial pressure in the brain). It is planned that this information gained will help develop dosing strategies that will achieve target concentrations that will successfully treat central nervous system infections in the future.

DETAILED DESCRIPTION:
Although relatively less frequent, Gram negative nosocomial meningitis and ventriculitis are observed in critical care settings, often associated with brain trauma, brain surgery, spinal fluid shunt after brain surgery, spinal abnormalities or severe urinary tract infections with bacteraemia. Gram negative meningitis is particularly challenging for treatment, when reduced susceptibility of some of the common etiologic bacteria is encountered (e.g. Acinetobacter baumannii, Pseudomonas aeruginosa, Enterobacter aerogenes). Furthermore, the presence of the blood brain barrier (BBB) has meant that the choice of systemic antibiotics is very restricted due to the limited ability of many antibiotics to achieve adequate concentrations in the cerebrospinal fluid (CSF). The poor CSF penetration may also contribute to an accelerated rate of the emergence of resistant pathogens in some patients/units. A significant proportion of Gram negative bacilli clinical isolates (from patients with meningitis) are resistant to broad spectrum antibiotics such as the third or later generation cephalosporins. With the wide spread use of these antibiotics, the incidence of resistant nosocomial infections has increased. Thus, there is an acute need for novel antibiotics that can achieve adequate concentrations in the CSF, while exhibiting an excellent spectrum of activity.

Ceftolozane/tazobactam is an emerging newly available antibiotic that has a broad spectrum of activity, and could be potentially useful in the management of Gram negative meningitis. As compared to other commonly used beta lactam antibiotics, it exhibits superior antibacterial activity against difficult to treat Gram negative organisms, such as Pseudomonas aeruginosa and Enterobacteriaceae spp. It is relatively stable against various resistance mechanisms encountered by other beta lactams, and may be useful in the treatment of multi-drug resistant (MDR) infections. However, data relating to CSF penetration is limited. In the critically ill, achieving adequate antibiotic exposure, especially against the high MIC of some Gram negatives (e.g. Pseudomonas), is difficult even in plasma, let alone in CSF for which a distribution barrier (i.e. BBB) exists. Thus, it is prudent to investigate the CSF pharmacokinetics of this new drug before it is used 'off label' by clinicians without supportive data.

This study will describe the plasma and CSF pharmacokinetics of a 3.0 g dose of ceftolozane/tazobactam in critically ill patients with an indwelling external ventricular drain (EVD). We will use a population pharmacokinetics approach to determine if altered dosing or alternative modes of administration, such as prolonged infusion, should be considered to improve plasma exposure. Given that direct administration into the CSF (e.g. intraventricular route) is not only invasive but also may risk neurotoxicity, pharmacokinetic studies should explore the extent of drug distribution into CSF with systemic administration. There is no clinical data on the CSF penetration of ceftolozane/tazobactam in critically ill patients at the moment, and as such, this is a highly valuable study.

Aim of the study is to describe the pharmacokinetics of a single dose of ceftolozane/tazobactam in the plasma and CSF of critically ill patients with an indwelling EVD.

The study investigators hypothesise:

The plasma PK of cefolozane/tazobactam may be altered in critically ill patients with an indwelling EVD.

The distribution of ceftolozane/tazobactam into the CSF may be impaired by the blood brain barrier.

ELIGIBILITY:
Inclusion Criteria:

Patients with any infection requiring treatment with ceftolozane/tazobactam and who have met the following criteria:

* Age >18 years
* The presence of an indwelling external ventricular drain (EVD) or requiring EVD insertion due to obstructive hydrocephalus/subarachnoid haemorrhage

Exclusion Criteria:

* Known or suspected allergy to penicillins and cephalosporins
* Pregnancy
* Receiving renal replacement therapy
* Glomerular filtration rate less than 10 mL/min
* Receiving piperacillin/tazobactam or having received piperacillin/tazobactam in the past 7 days before enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Roberts, PhD BPharm, Principal Investigator — Royal Brisbane and Womens Hospital
Locations (1):
- Royal Brisbane and Women's Hospital, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

RESULTS

PARTICIPANT FLOW:
Groups:
- Ceftolozane Tazobactam: Infected patients with external intraventricular drain will receive a single dose of Ceftolozane/ tazobactam (3000mg) over 1 hour and will undergo blood , csf and urine sampling at specific times over an 8 hour period.
  Ceftolozane/tazobactam: IV ceftolozane 2000mg /tazobactam 1000mg once only
Period: Overall Study
Arm/Group | Ceftolozane Tazobactam
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ceftolozane Tazobactam
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.5 [53.5 to 64.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 10
Weight [Median (Inter-Quartile Range); unit: kg] | 75 [65 to 87]
Serum Creatinine [Median (Inter-Quartile Range); unit: micro-mole/litre] | 48.5 [42.25 to 57.75]
Albumin [Median (Inter-Quartile Range); unit: g/L] | 24 [21.25 to 25.75]
Acute Physiology and Chronic Health Evaluation (APACHE) II [Median (Inter-Quartile Range); unit: units on a scale] — Acute Physiology and Chronic Health Evaluation II [APACHE II] score on ICU admission was calculated from 12 routine physiologic measurements using the standard approach. APACHE II score ranges from 1 to 71, with higher scores correlating with an increased risk of mortality. For a detailed description, please refer to Crit Care Med. 1985 Oct;13(10):818-29.
  units on a scale | 17.5 [14 to 22.5]

OUTCOME MEASURES:

1. Primary Outcome: Unbound Ceftolozane Exposure in the Plasma
Description: Unbound Ceftolozane Exposure in the plasma given by the area under the unbound concentration-time curve from time zero to infinity (AUC0-inf).
Time Frame: Samples collected from 0 to 8 hours post dose at "0, 1, 2,4,6, & 8 h post dose were use estimate area under the curve from time zero to infinity estimated by non-compartmental analysis
Measure: Median (Inter-Quartile Range); unit: mg*h/L
Arm/Group | Ceftolozane Tazobactam
Number analyzed (Participants) | 10
mg*h/L | 322.6 [182.7 to 413.9]

2. Primary Outcome: Unbound Tazobactam Exposure in the Plasma
Description: Unbound Tazobactam Exposure in the plasma given by the area under the unbound concentration-time curve from time zero to infinity (AUC0-inf).
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg*h/L
Arm/Group | Ceftolozane Tazobactam
Number analyzed (Participants) | 10
mg*h/L | 52.1 [35.7 to 79.6]

3. Primary Outcome: Unbound Ceftolozane Exposure in the CSF
Description: Unbound Ceftolozane Exposure in the CSF given by the area under the unbound concentration-time curve from time zero to infinity (AUC0-inf).
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg*h/L
Arm/Group | Ceftolozane Tazobactam
Number analyzed (Participants) | 10
mg*h/L | 30.2 [18.8 to 128.3]

4. Primary Outcome: Unbound Tazobactam Exposure in the CSF
Description: Unbound Tazobactam Exposure in the CSF given by the area under the unbound concentration-time curve from time zero to infinity (AUC0-inf).
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg*h/L
Arm/Group | Ceftolozane Tazobactam
Number analyzed (Participants) | 10
mg*h/L | 5.6 [1.6 to 24.4]

ADVERSE EVENTS:
Time Frame: The duration of the study enrolment up to 24 hours.
Arm/Group | Ceftolozane Tazobactam
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT03309657/Prot_SAP_000.pdf